CLINICAL TRIAL: NCT07290179
Title: Evaluating the Validity and Feasibility of a Smartwatch-based Eating Detection System to Passively and Automatically Detect Eating Events in Child-parent Dyads
Status: Not yet recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Hanim Diktas, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 2025-029
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Eating Behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Smartwatch and EMA-based eating behavior tracking — Participants (child-parent dyads) will wear a smartwatch on their dominant hand during a laboratory session and for three days in free-living conditions. In the lab, dyads will perform eating-related activities (e.g., eating with utensils, eating with hands, drinking) and non-eating activities (e.g., walking, writing, brushing teeth) while being video recorded for ground truth validation. Parents will receive a 20-minute training on using Ecological Momentary Assessment (EMA) prompts to record meal and snack times and will respond to EMA reminders during the free-living period. Adherence will be monitored through smartwatch wear time and EMA response rates.

SUMMARY:
This study will test the validity and feasibility of an smartwatch-based system to detect eating and drinking events in both laboratory and free-living conditions.

DETAILED DESCRIPTION:
The study will: 1) determine whether the smartwatch-based system accurately detects eating events in child-parent dyads in controlled settings and 2) evaluate the feasibility and practicality of passively detecting eating events in child-parent dyads over 3 days in free-living settings. The study will include two phases. During the laboratory visit, child-parent dyads will wear the smartwatch on their dominant hand and perform activities including eating gestures. These activities will be recorded with a video camera, and the videos will be coded for the ground truth times of eating. In the second phase of the study, child-parent dyads will continue wearing the smartwatch for 3 more days in free-living conditions. In the free-living period, parents will receive personalized Ecological Momentary Assessment (EMA) prompts reminding them to activate the smartwatch.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers (18-70 years) who have children aged 8-12 years
* Child is willing and able to wear smartwatch during school hours (have not restrictions in the school setting)

Exclusion Criteria:

* Any condition or circumstance that could impede study completion
* Child does not follow a regular eating pattern
* Child eats less than 1 meal and 1 snack in a day
* Child is restricted or allergic to the study foods
* Refusal or unable to use the smartwatch to collect data for the 3-day period in free - living conditions
* Parental refusal or unable to respond Ecological Momentary Assessment prompts

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A sample of 35 dyads (35 parents and their 8-12 years old children) will be recruited from the Baton Rouge, LA area.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy and Performance of Smartwatch-based Eating Detection System in Controlled Conditions | During the controlled laboratory session (Day 1).
  Accuracy and performance of smartwatch-based system for detecting eating and drinking events compared to video-coded ground truth during a controlled laboratory conditions. Metrics include:
  Precision (proportion of correctly detected eating events among all detected events), Recall/Sensitivity (proportion of actual eating events detected), Specificity (proportion of non-eating events correctly identified as non-eating) F1-score (harmonic mean of precision and recall), Overall accuracy (proportion of correct classification).
Adherence to Smartwatch Protocol | During the free-living phase (Days 2-4).
  Proportion of families meeting adherence criteria, defined as both parent and child wearing the smartwatch during eating on at least 2 of 3 days and the parent responding to ≥75% of EMA prompts related to smartwatch charging and app functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Hanim E Diktas, PhD, Principal Investigator — Pennington Biomedical Research Center